CLINICAL TRIAL: NCT04200586
Title: The Effects of SGLT Inhibition on Diabetic Cardiomyopathy
Brief Title: The Effects of SGLTi on Diabetic Cardiomyopathy
Acronym: SGLTi
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chung-Wah David SIU, Clinical Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version no.3
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Type2 Diabetes; Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Single-arm, observational
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dapagliflozin (Experimental): Dapagliflozin, one of the SGLT-2 inhibitors, will be prescribed to DM patients on clinical ground
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin, one of the SGLT-2 inhibitors, will be prescribed to DM patients on clinical ground.

SUMMARY:
Diabetic cardiomyopathy is associated with significant morbidity and mortality. It is considered as a cardiac muscle disorder secondary to diabetes mellitus (DM). Certain studies show the clinical benefit of SGLT-s inhibitors on reducing cardiovascular outcomes amongst patients with type II DM that go beyond the correction of hyperglycemic perse. Thus an observational imaging study is proposed to identify mechanistic insights of the drug group over cardiovascular events.

DETAILED DESCRIPTION:
Diabetic cardiomyopathy is defined as ventricular dysfunction in diabetic patients in the absence of coronary artery disease and hypertension. It is considered as a cardiac muscle disorder due to the metabolic consequences of DM characterized by left ventricular hypertrophy, left ventricular diastolic dysfunction (in the early stage), and/or systolic dysfunction. To date, there is no specific treatment proven effective for the condition due to the incomplete understanding of the pathogenesis.

Recent studies however prove the efficacy of SGLT-2 inhibitors on reducing the primary composite end point of cardiovascular outcomes including hospitalization for heart failure, cardiovascular death, and all-cause death amongst patients with type II DM. Such clinical benefit is apparently mainly stemmed from the reduction in heart failure related mortality and sudden cardiac death rather than the macro-vascular events such as myocardial infarct and stroke, suggesting addition benefits going beyond the correction of hyperglycemia perse. These studies thus raise the possibility that the drug may have direct effects on the myocardium that conferring the clinical benefit not related the modification of traditional risk factors such as glycemic control, lipid, blood pressure, and obesity.

A single-arm, observational cardiac magnetic resonance imaging study is proposed in type II diabetic patients before and 2 months after initiation of dapagliflozin. The aim is to identify mechanistic insights leading to the unexpected clinical benefit of SGLT inhibition.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* 40-90 years old
* HbA1c >= 6.5%
* history of heart failure with reduced ejection fraction
* indications for SGLT inhibition on clinical ground

Exclusion Criteria:

* angina pectoris or chest discomfort
* prior coronary artery bypass grafts
* coronary artery stenting within 6 months of study enrolment
* pervious myocardial infarct
* any contraindication for stress CMR testing
* renal impairment with eGFR <45ml/min/1.73m2
* limited life expectancy <5 years, for example due to pulmonary disease, cancer or
* significant hepatic failure
* contraindication to dapagliflozin or other SGLT2 inhibitors
* unable to take dapagliflozin
* patients currently on and SGLT2 inhibitor
* planned need for concomitant cardiac surgery or coronary intervention
* refusal or inability to sign an informed consent
* potential for on-compliance towards the requirements in the trial protocol (especially the medical treatment) or follow-up visits

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04-09 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in myocardial perfusion reserve index | 8-12 weeks
  Change in myocardial perfusion reserve index calculated from cardiac MRI

CONTACTS AND LOCATIONS:
Overall Officials: David Chung-Wah SIU, Prof, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong